CLINICAL TRIAL: NCT00712127
Title: Preventing Adverse Effects In Class II and Class III Obesity
Brief Title: Re-energize With Nutrition, Exercise and Weight Loss
Acronym: RENEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Bret Goodpaster, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0608088
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Body Fat; Exercise; Metabolic syndrome; Obesity; Nutrition; Physical Activity; Weight Loss
MeSH Terms: conditions — Obesity; Motor Activity; Metabolic Syndrome; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet and Exercise (Experimental): Diet and Exercise for Class II and Class III Obesity
  Interventions: Other: Diet and Exercise
- Diet and Exercise-Delayed (Experimental): Diet and Exercise-Delayed for 6 months for Class II and Class III Obesity
  Interventions: Other: Diet and Exercise-Delayed
- Control (No Intervention): Normal weight, overweight and Class I obesity

INTERVENTIONS:
Other: Diet and Exercise — The participants in this intervention will receive 12 months of weight loss through diet and exercise
  Arms: Diet and Exercise
Other: Diet and Exercise-Delayed — Participants in this intervention will receive six months of weight loss through diet followed by six months of diet and exercise
  Arms: Diet and Exercise-Delayed

SUMMARY:
The purpose of this project is to establish a Center of Excellence in Research on Obesity that will focus on severe obesity. The prevalence of severe obesity (i.e., Class 2 and 3 obesity; body mass index > 35 kg/m2 and 40 kg/m2) is increasing more rapidly than is overweight and Class 1 obesity. Treatment guidelines for severe obesity are uncertain.

Three novel hypotheses regarding the pathogenesis of severe obesity will be tested: a) using non-invasive methods to measure energy expenditure; b) conducting an annotated lipomic search for bio-markers of impaired fat oxidation; and c) examining the role of obesity-induced inflammation as a cause for leptin resistance. Responses will also be measured following intervention with diet and activity.

DETAILED DESCRIPTION:
SPECIFIC AIMS The first specific aim is to examine mechanisms for the pathogenesis of severe obesity.

Obesity is a heterogeneous and complex metabolic disorder. The pathogenesis of obesity remains obscure and it is unclear why some individuals are prone to severe obesity. It is also unclear why there are ethnic and racial differences for severe obesity. Many scientists postulate that metabolic vulnerabilities for obesity can be identified in the severely obese. The 1st specific aim examines the pathogenesis of severe obesity with three research protocols applied within the same cohort of research participants.

1. energy expenditure. Some prior studies indicate lower rates of resting energy expenditure (REE) in African-Americans, posing a metabolic risk for weight gain and resistance to weight loss. Other recent work highlights an important role for non-exercise activity thermogenesis (NEAT) in the pathogenesis of obesity. There are limited data addressing energy expenditure in severe obesity. In 120 severely obese adults (50% Class II and 50% Class III; with 50% African American participation), energy expenditure will be studied at baseline and after 6 months of intervention. The doubly-labeled water method will be used to measure total daily energy expenditure (TEE). Indirect calorimetry will be used to measure resting metabolic rate (RMR). Physical activity will be measured using light-weight, wearable monitors. NEAT will be calculated using these measurements. Comparisons will be between the groups with Class II and III obesity with further analysis for effects of ethnicity. These findings will be compared to data obtained in lean control subjects. The effect of intervention will be examined. This cohort will have a 1 year intensive behavioral weight loss intervention. Half of the volunteers will be randomized to a combined diet and exercise intervention (DE) , and the others will be randomized to diet intervention only for the initial 6 months, adding the exercise component at 6 months (DE-DELAY).
2. impaired capacity for fat oxidation. In these participants, a drop of blood will be obtained at baseline and 6 months, for a low-cost, high throughput, yet highly detailed tandem mass spectroscopy profile of plasma levels of acylcarnitines. Elevated levels will denote disorders of fatty acid oxidation and selective increase in specific acylcarnitine species will denote particular enzymatic loci of impairment. This aim derives from rapid recent progress in two parallel field of metabolic investigation. One of these is the field of "inborn errors of metabolism", a field generally applied to newborns and children. In this field there has been a rapid increase during the past decade in recognizing and delineating in-born errors of fatty acid oxidation. Profiling plasma levels of acylcarnitine species is a standard diagnostic approach. In obesity research, a strong body of data have been developed during the same interval that one of the key metabolic impairments is mitochondrial dysfunction and reduced capacity for fatty acid oxidation in skeletal muscle. Racial differences in muscle oxidative capacity have been reported, with lower values for oxidative capacity in AA women, characteristics postulated to be a metabolic risk factor for obesity. We propose inter-action of these two lines of investigation, exploring the utility of tandem mass spectroscopy screening for plasma acylcarnitines as a non-invasive probe of metabolic impairments in the severely obese.
3. leptin resistance. The third protocol to be used in this group of severely obese concerns a novel concept for leptin resistance. A decade ago, the discovery of leptin was pivotal in renewing scientific interest in obesity. Leptin modulates appetite and energy expenditure, two processes fundamental to weight regulation. Yet, treatment of obesity with leptin has failed to meet expectations. This has been attributed to "leptin resistance". This protocol will examine the role of serum leptin interacting proteins (SLIPs) that bind leptin as a factor contributing to leptin resistance. This line of basic science research indicates that one of the SLIPs is C-reactive protein (CRP) which suggests that low-grade inflammation, a metabolic complication of obesity related to risk for cardiovascular disease (CVD) may also contribute to the pathogenesis of obesity. There are common themes in these three protocols that form Specific Aim 1. Each addresses an aspect of the regulation of energy expenditure and fat oxidation. Each has the potential to identify novel bio-markers. Each project employs state-of-the-art analytical procedures, yet uses only minimally invasive sample collections. Finally, each will be carried out in the full research cohort of Phase 1, at baseline and during intervention, comparing metabolic effects of DE versus DE-DELAY. Though physical activity may be more important for weight loss maintenance than induction of weight loss, it has been found to increase capacity for fat oxidation more than weight loss induced by diet. It is from this latter perspective that we are interested in comparisons of DE and DE-DELAY at 6 months using these metabolic parameters.

The 2nd specific aim is to develop an effective intervention for the severely obese.

Axiomatic in the contemporary approaches to treatment of obesity is that clinically significant benefits are obtained with modest weight loss. This principle underlies the consensus recommendations for a weight loss target of 5 to 10% for overweight and obese individuals. The 2nd specific aim is to implement a behavioral dietary and physical activity intervention and assess whether this achieves a target weight loss at 1 year of ≥ 7% in Class II and Class III obese research participants. 120 adults, as described above, will have a 1 year intervention. Intervention to increase physical activity in the severely obese may be particularly challenging. Possibly this is easier after a period of weight loss. The staging of diet and physical activity (DE versus DEDELAY) will examine this.

The 3rd specific aim is to assess the effect of intervention on adverse health risks.

The medical rational for weight loss and physical activity is to improve health and ameliorate adverse effects of obesity. The 3rd specific aim is to assess the impact of intervention in the Phase 1 cohort. A panel of standardized clinical measurements, laboratory tests, and self-report instruments will be performed at baseline, 6 months and 1 year. We will examine: 1) traditional cardiovascular risk factors (e.g. hypertension, dyslipidemia, glucose and insulin, along with other endocrine measurements); 2) markers of inflammation, adipokines and cytokines; 3) body composition and regional distribution of adipose tissue; 4) functional status (a timed 400 meter corridor walk); 5) sub-clinical vascular disease (pulse wave velocity and carotid ultrasound); 7) health history and use of medications; and 8) demographic indices, social and neighborhood factors, quality of life, impact of obesity, and self-perception of body image and discrimination. One line of inquiry concerns the role of baseline characteristics in accounting for heterogeneity between individuals in adverse effects of severe obesity. The second line of inquiry is to assess the impact of intervention to change these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Overweight
* Age 30 to 55
* Able to walk 3 to 4 blocks
* Able to attend weekly meetings

Exclusion Criteria:

* Do not have diabetes
* Have not been in a weight loss program in the last year
* Have never had bariatric surgery or stomach bypass surgery
* Are not taking steroids or blood thinners
* Have no history of heart disease, heart attacks, heart surgery
* Have not had cancer in the past 5 years
* Are not pregnant, or haven't been in the past six months
* Are not currently nursing or planning to become pregnant in the next year
* Are not planning to move out of the area in the next year

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2006-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
This project addresses an important aspect of health disparity. The scientific inquiry as to causes of severe obesity seeks to determine if there is a differing metabolic disposition to obesity in AA compared to non-Hispanic White adults. | Twelve months

SECONDARY OUTCOMES:
To establish treatment guidelines for obesity. | Twelve Months

CONTACTS AND LOCATIONS:
Overall Officials: Bret H. Goodpaster, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Cheyney University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Fu CP, Ali H, Rachakonda VP, Oczypok EA, DeLany JP, Kershaw EE. The ZJU index is a powerful surrogate marker for NAFLD in severely obese North American women. PLoS One. 2019 Nov 26;14(11):e0224942. doi: 10.1371/journal.pone.0224942. eCollection 2019. PMID 31770380
- [Derived] Rachakonda V, Wills R, DeLany JP, Kershaw EE, Behari J. Differential Impact of Weight Loss on Nonalcoholic Fatty Liver Resolution in a North American Cohort with Obesity. Obesity (Silver Spring). 2017 Aug;25(8):1360-1368. doi: 10.1002/oby.21890. Epub 2017 Jun 12. PMID 28605159
- [Derived] Hames KC, Coen PM, King WC, Anthony SJ, Stefanovic-Racic M, Toledo FG, Lowery JB, Helbling NL, Dube JJ, DeLany JP, Jakicic JM, Goodpaster BH. Resting and exercise energy metabolism in weight-reduced adults with severe obesity. Obesity (Silver Spring). 2016 Jun;24(6):1290-8. doi: 10.1002/oby.21501. Epub 2016 Apr 30. PMID 27129892
- [Derived] Goodpaster BH, Delany JP, Otto AD, Kuller L, Vockley J, South-Paul JE, Thomas SB, Brown J, McTigue K, Hames KC, Lang W, Jakicic JM. Effects of diet and physical activity interventions on weight loss and cardiometabolic risk factors in severely obese adults: a randomized trial. JAMA. 2010 Oct 27;304(16):1795-802. doi: 10.1001/jama.2010.1505. Epub 2010 Oct 9. PMID 20935337